CLINICAL TRIAL: NCT06353516
Title: Evaluation of the Effect of Intravenous Anesthesia Versus Volatile Anesthesia on Blood-brain Barrier Permeability and Neuroinflammation Affecting Postoperative Cognitive Dysfunction in Elderly Patients: A Randomized Controlled Trial
Brief Title: The Effect of Intravenous Versus Volatile Anesthesia on Postoperative Cognitive Dysfunction in Elderly Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chung-Ang University Gwangmyeong Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Eun Jung Oh, Assistant Professor, Chung-Ang University Gwangmyeong Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2310-117-126
Record Dates: First submitted 2024-02-13; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: total intravenous anesthesia; inhaled gas anesthesia; blood-brain barrier permeability; neuroinflammation; delirium; postoperative cognitive dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications; Neuroinflammatory Diseases; Delirium | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Intervention Model Description: The participants are randomly assigned to total intravenous anesthesia group or inhaled gas anesthesia group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study is a double-blinded randomized controlled trial. The group assignment is conducted by the pre-generated random number table. The participant, investigator and the outcome assessor are blinded to the group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous Anesthesia (Active Comparator): The anesthesia is maintained with intravenous anesthetics
  Interventions: Drug: Propofol
- Inhaled Gas Anesthesia (Sham Comparator): The anesthesia is maintained with inhaled gas anesthetics
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — delivered via intravenous route
  Arms: Intravenous Anesthesia
Drug: Sevoflurane — delivered via inhalation route
  Arms: Inhaled Gas Anesthesia

SUMMARY:
The goal of this clinical trial is to compare the permeability of blood-brain barrier between the intravenous anesthesia group and the inhalation gas anesthesia group in the elderly patients undergoing surgery. The main questions it aims to answer are:

* [Is the permeability of blood-brain barrier between the intravenous anesthesia group and the inhalation gas anesthesia group in the elderly patients different?]
* [Is the incidence of postoperative cognitive dysfunction between the intravenous anesthesia group and the inhalation gas anesthesia group different?] Participants will be anesthetized with different categories of anesthetics.

  * Intravenous anesthetics
  * Inhalation gas anesthetics

DETAILED DESCRIPTION:
This clinical trial targets patients aged 60 years or older with American Society of Anesthesiologists physical status (ASA) 1 to 3 who undergo surgery under general anesthesia at our hospital. Before entering the operating room, patients are randomly assigned to the intravenous anesthesia group and the inhalation gas anesthesia group. The intravenous anesthesia group uses propofol for anesthesia, and the inhalation gas anesthesia group uses sevoflurane. A 3 mL blood sample is collected four times: before surgery, at the end of surgery, 4 hours after surgery, and 1st day after surgery. All blood samples will be immediately transferred to the department of Laboratory medicine and stored at -80 degree. Pre-scheduled tests to determine the brain-blood barrier permeability and inflammatory cytokines will be conducted after the recruitment of all samples. In addition, for patients scheduled to be transferred to the intensive care unit (ICU) after surgery among the study subjects, a 3 mL of cerebrospinal fluid sample is collected two times: before surgery, and at the end of surgery. The same preservation protocol will be applied to the cerebrospinal fluid samples. All study subjects will be monitored for postoperative delirium daily for up to 7 days after surgery or until discharge. Cognitive function is assessed using telephone version of the Montreal Cognitive Assessment (T-MOCA) before surgery and 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* age equal to or older than 60
* american Society of Anesthesiologists (ASA) grade I to III
* general anesthesia longer than 2 hours

Exclusion Criteria:

* history of dementia
* history of schizophrenia, epilepsy, or Parkinson's disease
* history of stroke or craniectomy
* patient denial

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of serum S100B levels | before surgery, at the end of surgery, 4 hours after surgery, 1st day after surgery
  Levels of S100B will be obtained from venous blood samples collected before surgery, at the end of surgery, 4 hours after surgery, and 1st day after surgery.

SECONDARY OUTCOMES:
Incidence of Delirium | during 7 postoperative days or until discharge if the postoperative hospital stay is shorter than 7 days
  Investigators will investigate the occurrence of Delirium using CAM or CAM-ICU (in case of ICU admission). during 7 postoperative days or until discharge if the postoperative hospital stay is shorter than 7 days.
Incidence of Postoperative Cognitive Dysfunction | before surgery, 3 months after surgery
  The T-MOCA is a validated cognitive function test. The investigators will investigate changes in T-MOCA between baseline and 3 months after surgery.
Concentration of serum albumin | before surgery, at the end of surgery, 4 hours after surgery, 1st day after surgery
  Levels of albumin will be obtained from venous blood samples collected before surgery, at the end of surgery, 4 hours after surgery, and 1st day after surgery.
Concentration of serum CRP | before surgery, at the end of surgery, 4 hours after surgery, 1st day after surgery
  Levels of CRP will be obtained from venous blood samples collected before surgery, at the end of surgery, 4 hours after surgery, and 1st day after surgery.
Concentration of serum IL6 levels | before surgery, at the end of surgery, 4 hours after surgery, 1st day after surgery
  Levels of IL6 will be obtained from venous blood samples collected before surgery, at the end of surgery, 4 hours after surgery, and 1st day after surgery.
Concentration of serum TNFα levels | before surgery, at the end of surgery, 4 hours after surgery, 1st day after surgery
  Levels of TNFα will be obtained from venous blood samples collected before surgery, at the end of surgery, 4 hours after surgery, and 1st day after surgery.
Concentration of cerebrospinal fluid (CSF) albumin | Within 24 hour before surgery, at the end of surgery
  (in case of schedulled ICU admission) Levels of albumin will be obtained from CSF samples collected before surgery, at the end of surgery in case of schedulled ICU admission.

CONTACTS AND LOCATIONS:
Overall Officials: Eun Jung Oh, M.D., Ph.D., Study Director — Chung-Ang University Gwangmyeong Hospital
Locations (1):
- Chung-Ang University Gwangmyeong Hospital, Gwangmyeong, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlies the results of this study will be made available upon reasonable request, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Data will be available to researchers who provide a methodologically sound proposal to the corresponding author of the article. To gain access, data requestors will need to sign a data access agreement.